CLINICAL TRIAL: NCT03390270
Title: Rational Coronary Care Unit Triage for Stable Patients With NSTEMI: Evaluating the Safety and Costs of a Risk Score-based Triaging System
Brief Title: Risk-score Based ICU Triage
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00080891
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Non-ST Elevation Myocardial Infarction (nSTEMI)
Keywords: intensive care units; critical care; risk assessment; electronic health records
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with NSTEMI: All patients admitted to Duke University Hospital with an NSTEMI
  Interventions: Other: Admission with NSTEMI

INTERVENTIONS:
Other: Admission with NSTEMI — All patients admitted to Duke University Hospital with an NSTEMI

SUMMARY:
The investigators have created a new risk score that predicts whether initially stable patients with myocardial infarctions (heart attacks) will require intensive care while they are in the hospital. To evaluate how well this risk score works, the investigators plan to calculate this risk score for every patient that comes to the hospital with a heart attack, provide the risk score to the emergency room doctor treating the patient, and determine whether each patient required intensive care while they were in the hospital. The investigators will then evaluate whether giving emergency room doctors access to this risk score reduced costs of taking care of heart attack patients compared with previous years.

DETAILED DESCRIPTION:
Multiple recent studies have demonstrated considerable between-hospital variability in ICU utilization for stable patients with NSTEMI and a lack of association between higher hospital-level ICU utilization and short-term mortality. Moreover, severity of illness, as measured by a traditional in-hospital mortality risk score, has only a trivial correlation with ICU utilization. A minority of initially stable patients with NSTEMI (~15%) deteriorates clinically while hospitalized and requires ICU care for management of cardiac arrest, shock, arrhythmias requiring pacing, stroke, or respiratory failure. Across a variety of conditions outcomes are better when patients are admitted directly to the ICU from the emergency department (ED) rather than transferred in after admission. However, the cost of caring for patients in the ICU is substantially more than the cost of caring for these patients in a non-ICU environment. Furthermore, treating patients that do not require intensive care in the ICU exposes them to unnecessary risks of ICU care, including medication errors, adverse procedural outcomes, delirium, and excessive noise. Reducing ICU utilization for stable patients with NSTEMI may reduce costs and improve patient satisfaction.

Using data from a nationally-representative registry enrolling patients with acute MI, the investigators developed the ACTION ICU risk score. Incorporating demographic, clinical, and laboratory data obtained routinely in the ED work-up of patients with suspected acute MI, the ACTION ICU risk score calculates the risk of in-hospital complications mandating ICU care for initially stable patients with NSTEMI. Complications mandating ICU care were defined as death, shock (cardiogenic or otherwise), cardiac arrest, high degree heart block requiring pacemaker placement, respiratory failure, or stroke. The risk score's c-statistic was 0.72, indicating good discrimination. Importantly, it identified > 50% of patients as being at < 10% risk of in-hospital complications mandating ICU care.

However, the clinical and financial implications of using this score to guide ICU triage in routine clinical practice are unknown, and the risk score has not been prospectively validated.

The investigators will create a calculator for the electronic health record that automatically calculates the ACTION ICU risk score for all patients with NSTEMI, as identified by their initial troponin value. Once the score is calculated, it will provide the score, and the patient's risk of clinical deterioration to the ED physician, along with a recommendation for where patients at that risk should be treated. The ED physician, working with the cardiologist on call, will then decide where the patient should be treated.

After one year, each patient for whom the score was calculated will be identified by a query of the electronic medical record. From the electronic medical record, the investigators will identify whether the patient was initially admitted to the ICU or to a non-ICU unit, whether the patient was transferred to the ICU during their hospital course, and whether the patient had clinical complications mandating ICU care (death, shock, cardiac arrest, heart block requiring pacemaker, stroke, or respiratory failure). The investigators will also compare total hospital costs for caring for NSTEMI patients before and after roll-out of the ACTION ICU score electronic medical record plug-in. Study completion will be defined by the last date of data extracted from the medical records for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Presents to DUMC with elevated cardiac troponin
* Identified by ED physician as having myocardial infarction

Exclusion Criteria:

* ST segment elevation myocardial infarction
* Hemodynamically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Duke University Medical Center Emergency Department with elevated cardiac troponin
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Hospital cost in dollars | 1 year
  Cost of caring for NSTEMI patients at Duke University Hospital in the 1 year prior to roll-out of the risk score versus the 1 year after

SECONDARY OUTCOMES:
ICU transfer | 30 days
  Whether a patient initially admitted to a non-ICU setting is transferred to the ICU during the index hospitalization
Development of complications mandating ICU care during the index hospitalization | 30 days
  Composite of death or development of shock, cardiac arrest, heart block requiring treatment, stroke, or respiratory failure (as identified by billing codes)
Death during the index hospitalization | 30 days
  Element of composite of "complications mandating ICU care"
Shock during the index hospitalization | 30 days
  Element of composite of "complications mandating ICU care"; defined by billing codes
Cardiac arrest during the index hospitalization | 30 days
  Element of composite of "complications mandating ICU care"; defined by billing codes
Heart block requiring treatment during the index hospitalization | 30 days
  Element of composite of "complications mandating ICU care"; defined by billing codes
Stroke during the index hospitalization | 30 days
  Element of composite of "complications mandating ICU care"; defined by billing codes
Respiratory failure during the index hospitalization | 30 days
  Element of composite of "complications mandating ICU care"; defined by billing codes

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fanaroff, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No